CLINICAL TRIAL: NCT03950258
Title: Endovascular Management of Pediatric Intracranial Arteriovenous Shunts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, osama mahmoud ahmed ramadan, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endovascular in pediatric
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Arteriovenous Malformations; Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Malformations; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endovascular embolization (Experimental): patients under the age of 18 years with arteriovenous shunts manifested by systemic or neurological manifestations will undergo endovascular embolization
  Interventions: Procedure: endovascular embolization

INTERVENTIONS:
Procedure: endovascular embolization — Transarterial embolization is done for patients with arteriovenous shunts as via transfemoral access using flow-guided microcatheter and an embolic agent is injected.

SUMMARY:
* Review the outcomes of the Endovascular management of pediatric intracranial arteriovenous shunts.
* Give an effective treatment for pediatric intracranial arteriovenous shunts and can detect the best method could be used and assess safety and efficacy of different endovascular techniques in treatment of different AV shunts.
* Improve the outcome of these patients and decease rate of recurrence and complications.

DETAILED DESCRIPTION:
Intracranial arteriovenous shunts (ICAVS) in young children are characterized by frequent high-flow fistulas. In association with high-flow fistulas and the physiological condition of the developing brain and heart, each ICAVS type tends to present at a certain age with unique symptoms.

Vein of Galen aneurysmal malformation (VGAM) and dural sinus malformation with arteriovenous (AV) shunt tend to present in the neonate with high output cardiac failure. In infancy, VGAM, pial arteriovenous fistula (AVF) and infantile dural AVF (DAVF) tend to present with hydrodynamic disorder such as macrocephaly, ventriculomegaly, prominent facial veins, and developmental delay.

Pial AVF, AV malformation, and infantile DAVF can present with focal neurological signs such as seizure or hemorrhage at older ages they are in the subpial space, as opposed to VGAM or DAVF, which are extrapial in location and tend to present with systemic symptoms .

Endovascular treatment is currently the first choice of treatment for most pediatric ICAVS. The treatment goal should be defined on a patient-by-patient basis, according to the unique physiological condition of the child.

ELIGIBILITY:
Inclusion Criteria:

* 1- clinical manifestation of AV shunt according to the pathology with radiological diagnosis by CT angiography or MRA 2- patient must be under 18 years old

Exclusion Criteria:

1. Any patient above 18 years old
2. Asymptomatic patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Independent clinical outcome changes | within one week after treatment
  The changes in clinical condition of the patients will be assessed before and after treatment using modified Rankin scale, as the scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Radiological outcome: | Immediate post treatment and at 6 and 12 months post treatment
  CT angiography or MR angiography will be done to show complete or in complete occlusion of the AV shunt

CONTACTS AND LOCATIONS:
Overall Officials: Osama Ramadan, master, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No